CLINICAL TRIAL: NCT02603757
Title: Prospective Pilot Study to Assess the Effectiveness of Vitamin D Supplementation for Patients Requiring Chemotherapy for Stage III Colorectal Cancer
Brief Title: Effectiveness of High Dose Vitamin D Supplementation in Stage III Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Eric Anderson, Principal Investigator, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D & Colorectal Cancer
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Vitamin D
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Standard-dose of 2,000 IU Vitamin D3, daily
  Interventions: Dietary Supplement: cholecalciferol
- Group B (Experimental): Higher-dose of 50,000 IU of Vitamin D3, weekly
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 2,000 IU of Vitamin D3 daily and 50,000 IU Vitamin D3 daily
  Other Names: Vitamin D3

SUMMARY:
This is a pilot study to test whether there is an association between baseline Vitamin D levels, Vitamin D supplementation and survival in patients with stage III colon and stage II/III rectal cancer receiving chemotherapy. 70 patients with colon stage III or rectal stage II or III cancer that require chemotherapy will be screened and 60 patients will be enrolled. Patients will be randomized to standard dose (2000 IU daily) or high-dose (50,000 IU weekly) Vitamin D supplementation for 1 year after initiation of chemotherapy. Patients' Vitamin D levels will be checked throughout supplementation then followed for 5 years with occasional Vitamin D testing and surveying in order to collect information on recurrence and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Willing to stop herbal medications as directed by physician
* Willing to stop current supplemental Vitamin D (Multivitamin with Vitamin D component is acceptable)
* Willing to travel to Legacy Health/OHSU facility if necessary
* Agree to attend study visits outside of standard of care visits, if necessary
* Diagnosed with stage III colon or stage II/III rectal cancer that will receive neoadjuvant or adjuvant chemotherapy but have not yet started
* Baseline serum Vitamin D level below 52 ng/ml

Exclusion Criteria:

* ≤ 18 years of age
* Colon cancer stages I-II and IV or Rectal cancer stage I or IV
* Patients who do not undergo chemotherapy
* Patients with prior chemotherapy for this cancer
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cancer, or other cancer for which the patient has been disease-free for > 3 years
* Unable to comply with protocol
* Unable to provide written informed consent
* Unwilling or unable to stop oral supplemental Vitamin D
* Patients taking high-dose Vitamin D supplementation (50,000 IU weekly) prior to enrollment
* Patients with Vitamin D levels above 52 ng/ml at baseline testing
* Patients with hypercalcemia and/or any condition resulting in malabsorption
* Investigator does not believe study participation, for any reason, is in the best interest of the patient

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Increase in serum Vitamin D3 level during chemotherapy in the active supplementation group compared to the control group. | 1 year

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | 5 years
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Anderson, MD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Legacy Meridian Park Medical Center, Tualatin, Oregon

REFERENCES:
- [Background] Fiscella K, Winters P, Tancredi D, Hendren S, Franks P. Racial disparity in death from colorectal cancer: does vitamin D deficiency contribute? Cancer. 2011 Mar 1;117(5):1061-9. doi: 10.1002/cncr.25647. Epub 2010 Oct 13. PMID 20945439
- [Background] Zgaga L, Theodoratou E, Farrington SM, Din FV, Ooi LY, Glodzik D, Johnston S, Tenesa A, Campbell H, Dunlop MG. Plasma vitamin D concentration influences survival outcome after a diagnosis of colorectal cancer. J Clin Oncol. 2014 Aug 10;32(23):2430-9. doi: 10.1200/JCO.2013.54.5947. Epub 2014 Jul 7. PMID 25002714
- [Background] Ng K, Sargent DJ, Goldberg RM, Meyerhardt JA, Green EM, Pitot HC, Hollis BW, Pollak MN, Fuchs CS. Vitamin D status in patients with stage IV colorectal cancer: findings from Intergroup trial N9741. J Clin Oncol. 2011 Apr 20;29(12):1599-606. doi: 10.1200/JCO.2010.31.7255. Epub 2011 Mar 21. PMID 21422438
- [Background] Brunner RL, Wactawski-Wende J, Caan BJ, Cochrane BB, Chlebowski RT, Gass ML, Jacobs ET, LaCroix AZ, Lane D, Larson J, Margolis KL, Millen AE, Sarto GE, Vitolins MZ, Wallace RB. The effect of calcium plus vitamin D on risk for invasive cancer: results of the Women's Health Initiative (WHI) calcium plus vitamin D randomized clinical trial. Nutr Cancer. 2011;63(6):827-41. doi: 10.1080/01635581.2011.594208. Epub 2011 Jul 20. PMID 21774589
- [Background] Fakih MG, Andrews C, McMahon J, Muindi JR. A prospective clinical trial of cholecalciferol 2000 IU/day in colorectal cancer patients: evidence of a chemotherapy-response interaction. Anticancer Res. 2012 Apr;32(4):1333-8. PMID 22493367
- [Background] Fedirko V, Bostick RM, Flanders WD, Long Q, Shaukat A, Rutherford RE, Daniel CR, Cohen V, Dash C. Effects of vitamin D and calcium supplementation on markers of apoptosis in normal colon mucosa: a randomized, double-blind, placebo-controlled clinical trial. Cancer Prev Res (Phila). 2009 Mar;2(3):213-23. doi: 10.1158/1940-6207.CAPR-08-0157. Epub 2009 Mar 3. PMID 19258546
- [Background] Fernandez-Garcia NI, Palmer HG, Garcia M, Gonzalez-Martin A, del Rio M, Barettino D, Volpert O, Munoz A, Jimenez B. 1alpha,25-Dihydroxyvitamin D3 regulates the expression of Id1 and Id2 genes and the angiogenic phenotype of human colon carcinoma cells. Oncogene. 2005 Sep 29;24(43):6533-44. doi: 10.1038/sj.onc.1208801. PMID 16007183
- [Background] Fedirko V, Bostick RM, Long Q, Flanders WD, McCullough ML, Sidelnikov E, Daniel CR, Rutherford RE, Shaukat A. Effects of supplemental vitamin D and calcium on oxidative DNA damage marker in normal colorectal mucosa: a randomized clinical trial. Cancer Epidemiol Biomarkers Prev. 2010 Jan;19(1):280-91. doi: 10.1158/1055-9965.EPI-09-0448. PMID 20056649
- [Background] Bee CR, Sheerin DV, Wuest TK, Fitzpatrick DC. Serum vitamin D levels in orthopaedic trauma patients living in the northwestern United States. J Orthop Trauma. 2013 May;27(5):e103-6. doi: 10.1097/BOT.0b013e31825cf8fb. PMID 22576645
- [Background] Morgan SL, Weinsier RL. Fundamentals of clinical nutrition, Mosby, St. Louis 1998. p.3